CLINICAL TRIAL: NCT05939180
Title: Study of the Efficacy and Safety of Venetoclax Plus Azacytidine Versus Daunorubicin Plus Cytarabine in Adult Acute Myeloid Leukemia (AML) Patients With Adverse Risk Features
Brief Title: VA vs DA for Newly Diagnosed Hig-risk AML
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Victor AML-1
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2023-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: Adverse risk, newly diagnosed, induction therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine; Daunorubicin; Cytarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VA regimen (Experimental): VA regimen: azacytidine and venetoclax
  Interventions: Drug: Venetoclax Oral Tablet
- DA regimen (Active Comparator): DA regimen: daunorubicin and cytarabine
  Interventions: Drug: Daunorubicin

INTERVENTIONS:
Drug: Venetoclax Oral Tablet — VA regimen: azacytidine, 75mg/m2, subcutaneously, on days 1-7; venetoclax, orally, once a day, 100mg, d1; 200mg, d2; 400mg, days 3-28.
  Other Names: venetoclax plus azacytidine
  Arms: VA regimen
Drug: Daunorubicin — DA regimen: daunorubicin (60mg/m2) on days 1-3, intraveneously injection, and cytarabine (100mg/m2) on days 1-7, intraveneously injection, for 1 cycle.
  Other Names: daunorubicin plus cytarabine
  Arms: DA regimen

SUMMARY:
This is an open-label, multicenter, phase 2b, randomized study aiming to compare the efficacy and safety of venetoclax plus azacytidine Versus daunorubicin plus cytarabine (conventional 7+3 regimen) in adult acute myeloid leukemia (AML) patients with adverse risk featuress. Participants will be 1:1 randomly assigned to the VA and DA groups. Once remission was achieved, consolidated chemotherapy will be performed and allogeneic hematopoietic stem cell transplantation is strongly recommended. After completion of the study intervention, participants will be followed-up every 1 to 2 months for up to 2 years.

DETAILED DESCRIPTION:
This is an open-label, multicenter, phase 2b, randomized study aiming to compare the efficacy and safety of venetoclax plus azacytidine Versus daunorubicin plus cytarabine (conventional 7+3 regimen) in adult acute myeloid leukemia (AML) patients with adverse risk featuress. Newly diagnosed AML patients with adverse risk features according to 2022 European Leukemia Net risk stratification will be enrolled. In the study, a novel second generation targeted sequencing panel for the fast screening of adverse mutations with 72-hours after the bone marrow samples will be utilized. Randomized participants will receive induction treatment . Participants will be 1:1 randomly assigned to the VA and DA groups. VA regimen comprises of azacytidine, 75mg/m2, subcutaneously, on days 1-7; venetoclax, orally, once a day, 100mg, d1; 200mg, d2; 400mg, days 3-28. DA regimen comprises of daunorubicin (60mg/m2) on days 1-3, intraveneously injection, and cytarabine (100mg/m2) on days 1-7, intraveneously injection, for 1 cycle. Once remission was achieved, consolidated chemotherapy will be performed and allogeneic hematopoietic stem cell transplantation is strongly recommended. After completion of the study intervention, participants will be followed-up every 1 to 2 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: female or male.
2. Age:18-64 years old.
3. Patients with newly diagnosed AML according to the WHO 2022 classification.
4. AML patients with adverse risk features according to the 2022 European Leukemia Net risk stratification.
5. Untreated AML (hydroxyurea, and low dose cytarabine with cummulative dose <1.0g are permitted).
6. ECOG: 0-2.
7. Adequate liver function: Total bilirubin ≤ 1.5×upper limit of normal (ULN); aspartate aminotransferase (AST) ≤3×ULN (liver infiltration of leukemia: ≤5×ULN); alanine aminotransferase (ALT)≤3×ULN (liver infiltration of leukemia: ≤5×ULN) .
8. Adequate Renal function: Ccr (Creatinine Clearance Rate) ≥30 ml/min.
9. Be able to understand and be willing to participate in the study. Be able to provide written informed consent.

Exclusion Criteria:

1. Patients with acute promyeloid leukemia.
2. AML with central nervous system infiltration.
3. Patients diagnosed with myeloid sarcoma.
4. Patients have AML secondary to MDS and previously been treated with hypomethylating agents.
5. Patients with active infection, which is considered as uncontrollable by the investigator.
6. Patients with active hepatitis B, hepatitis C and HIV infection.
7. Patients with heart failure (grade 3-4);
8. Patients who are pregnant or breastfeeding.
9. Patients who refused to be enrolled in the study. Patients who are considered as ineligible for the enrollment by the investigators.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Composite complete remission (CRc) after one course of induction therapy | From randomization to the end of the first course of induction therapy (within 28 days)
  Rates of complete remission plus complete remission with incomplete blood cell rates of complete remission or complete remission with incomplete marrow recovery

SECONDARY OUTCOMES:
DOR: duration of remission | 2 years
  Time between the first remission and relapse
EFS：event-free survival | 2 years
  time from the date of enrollment to treatment failure, relapse, death from any cause or the last follow-up
OS: overall survival | 2 years
  time from the date of enrollment to death from any cause or the last follow-up
Volume of infused blood products | Within 60 days after randomization
  The volume of infused blood products during the induction treatment.
AE | Within 60 days after randomization
  Adverse events during the induction treatment.
Composite complete remission (CRc) after two courses of induction therapy | From randomization to the end one and two courses of induction therapy (within 60 days)
  complete remission or complete remission with incomplete marrow recovery

CONTACTS AND LOCATIONS:
Overall Officials: Su-ning Chen, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (2):
- China (2):
  - The First Affiliated Hospital of Soochow University, Jiangsu Institute of Hematology, Suzhou, Jiangsu
  - Ethical Committee of the First Affliated Hospital of Soochow University, Suzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No